CLINICAL TRIAL: NCT03046173
Title: Osteogenic Effects of Concentrated Growth Factors Applied in Maxillary Sinus Floor Elevation Via a Lateral Window Approach With Simultaneous Implant Placement: a Single-center Randomized Controlled Trial
Brief Title: Concentrated Growth Factors Applied in Maxillary Sinus Floor Elevation Via a Lateral Window Approach
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Deyang Stomatological Hospital (Other)
Responsible Party: Principal Investigator, Yang Cheng, Attending Physician, Deyang Stomatological Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DeyangSH_001
Record Dates: First submitted 2017-01-16; First posted 2017-02-08 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2017-02

CONDITIONS: Maxillary Sinus Disease
MeSH Terms: interventions — Durapatite

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- the experimental group (Experimental): These patients were randomly assigned to receive concentrated growth factors, hydroxyapatite and autogenous bone at bone defect sites in the experimental group.
  Interventions: Other: concentrated growth factors
- the control group (Experimental): These patients were randomly assigned to receive hydroxyapatite and autogenous bone at bone defect sites in the control group.
  Interventions: Other: hydroxyapatite and autogenous bone

INTERVENTIONS:
Other: concentrated growth factors — These patients were randomly assigned to receive concentrated growth factors, hydroxyapatite and autogenous bone at bone defect sites in the experimental group.
  Arms: the experimental group
Other: hydroxyapatite and autogenous bone — These patients were randomly assigned to receive hydroxyapatite and autogenous bone at bone defect sites in the control group.
  Arms: the control group

SUMMARY:
To investigate the effects of concentrated growth factors applied in maxillary sinus floor elevation via a lateral window approach with simultaneous implant placement on repair of bone defects and new bone formation.

DETAILED DESCRIPTION:
Maxillary sinus floor elevation via a lateral window approach is the most effective method of overcoming the shortage of bone mass deficiency in atrophic maxillary posterior region. Bone transplantation is considered to be a prerequisite for the success of maxillary sinus floor elevation. Platelet-rich plasma and platelet-rich fibrin have been used to accelerate bone formation, regeneration, and repair. However, few in-depth studies are reported on the effects of concentrated growth factors on new bone formation.

ELIGIBILITY:
Inclusion Criteria:

* Loss of one or more maxillary molars in the posterior maxillary region
* Occlusogingival distance of > 4 mm
* Residual bone height of 2-5 mm in the posterior maxillary region, no obvious maxillary sinus separation
* No problems with the lungs, heart, or brain
* Normal liver and kidney function
* Normal coagulation function
* Adequate prosthetic space
* No history of bruxism or temporomandibular joint disorders
* No tumors, cysts and polyps in maxillary sinus
* No acute or chronic maxillary sinusitis
* No acute periodontitis
* No oral mucosal disease
* Age 20-45 years
* Able to tolerate the stress of anesthesia and surgery

Exclusion Criteria:

* Residual bone height of < 1 mm in the posterior maxillary region or presence of maxillary sinus mucosa rupture
* Poor control of complex periodontal disease
* Local inflammation or poor oral hygiene
* Poorly treated maxillary disease
* With severe bruxism
* With temporomandibular joint disorders
* Alcohol consumption and cigarette smoking (20 cigarettes/d)
* Have a history of chemotherapy and radiation therapy in face and neck
* Pregnant
* With coagulation disorders
* With autoimmune disease
* With severe osteoporosis
* With acute maxillary sinusitis
* Unable to tolerate simple surgery because of systemic diseases including severe diabetes mellitus and heart disease
* Unable to provide informed consent

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2014-05; Primary Completion 2016-01 (Actual); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Excellent and good rate of bone repair | changes of month 1, month 3 and month 6 after surgery
  X-ray examination was performed to evaluate bone repair as per excellent and good rate.

SECONDARY OUTCOMES:
Bone density at bone defect sites | changes of month 1, month 3 and month 6 after surgery
  The thickness of the cortical bone at the defect sites was measured using a dental cone beam CT scanner to reflect bone density.

CONTACTS AND LOCATIONS:
Overall Officials: Min Liu, MD, Principal Investigator — Deyang Stomatological Hospital

IPD SHARING:
Plan to Share IPD: Undecided